CLINICAL TRIAL: NCT04019288
Title: Randomized Phase I/II Study of AVB-S6-500 in Combination With Durvalumab (MEDI4736) in Patients With Platinum-Resistant, Recurrent Epithelial Ovarian Cancer
Brief Title: AVB-S6-500 and Durvalumab in Treating Patients With Platinum-Resistant or Recurrent Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI Request
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Aravive Biologics Inc (Unknown); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0149; NCI-2019-02580 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0149 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Platinum-Resistant Fallopian Tube Carcinoma; Platinum-Resistant Ovarian Carcinoma; Platinum-Resistant Primary Peritoneal Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Refractory Fallopian Tube Carcinoma; Refractory Ovarian Carcinoma; Refractory Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — AVB-500 fusion protein; durvalumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (batiraxcept, durvalumab) (Experimental): Patients receive batiraxcept IV over 60 minutes on days 1, 15, and 29 of cycle 0, and on days 1 and 15 of subsequent cycles. Beginning cycle 1, patients also receive durvalumab IV over 60 minutes on day 1. Cycle 0 continues for 6 weeks and subsequent cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Batiraxcept; Biological: Durvalumab
- Arm II (durvalumab, batiraxcept) (Experimental): Patients receive durvalumab IV over 60 minutes on days 1 and 22 of cycle 0 and on day 1 of subsequent cycles. Beginning cycle 1, patients also receive batiraxcept IV over 60 minutes on days 1 and 15. Cycle 0 continues for 6 weeks and subsequent cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Batiraxcept; Biological: Durvalumab

INTERVENTIONS:
Drug: Batiraxcept — Given IV
  Other Names: Anti-AXL Fusion Protein AVB-S6-500; AVB S6 500; AVB-500; AVB-S6-500; AVBS6500; AXL Fc Fusion Protein AVB-S6-500; RUGA-S6
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736

SUMMARY:
This trial studies the side effects and best dose of AVB-S6-500 when given together with durvalumab in treating patients with ovarian, fallopian tube, or primary peritoneal cancer that is resistant to platinum therapy or has come back. Immunotherapy with AVB-S6-500 and durvalumab, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine toxicity profile of the combination of batiraxcept (AVB-S6-500) and durvalumab therapy.

SECONDARY OBJECTIVES:

I. To estimate objective response rate to combination AVB-S6-500 and durvalumab therapy.

II. To estimate the median immune-related progression free survival (irPFS) as well as overall survival (OS) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 after treatment with combination durvalumab and AVB-S6-500.

III. To investigate molecular and immunological changes associated with the combination of AVB-S6-500 and durvalumab; specifically to describe changes in T cell populations (including but not limited to CD3, CD8, CD4, FOXP3) and cell proliferation, as well as report changes in the proportion of macrophage phenotypes M1 and M2 (with phenotypic markers potentially including arginase1, CD11b, PDL-1, and CD206).

EXPLORATORY OBJECTIVES:

I. To evaluate blood and tissue based biomarkers for immune related adverse events and disease progression.

II. To investigate impact and possible sensitization of pretreatment with AVB-S6-500 monotherapy on subsequent combination of durvalumab and AVB-S6-500.

III. To evaluate for molecular and immunologic differences between pre-treatment with single agent AVB-S6-500 as compared to durvalumab.

OUTLINE: This is a phase I, dose-escalation of batiraxcept, followed by a phase II study. In Phase I, patients receive both batiraxcept (intravenously [IV] over 60 minutes on days 1 and 15) and durvalumab (IV over 60 minutes on day 1) every cycle.

In Phase II, patients are randomized to 1 of 2 arms.

ARM I: Patients receive batiraxcept IV over 60 minutes on days 1, 15, and 29 of cycle 0, and on days 1 and 15 of subsequent cycles. Beginning cycle 1, patients also receive durvalumab IV over 60 minutes on day 1. Cycle 0 continues for 6 weeks and subsequent cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive durvalumab IV over 60 minutes on days 1 and 22 of cycle 0 and on day 1 of subsequent cycles. Beginning cycle 1, patients also receive batiraxcept IV over 60 minutes on days 1 and 15. Cycle 0 continues for 6 weeks and subsequent cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 weeks for at least 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide signed informed consent
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
* Histology (reviewed at MD Anderson Cancer Center [MDACC]) showing recurrent high grade epithelial ovarian, peritoneal, or fallopian tube cancer
* Platinum resistant or refractory disease as defined by progression of disease on a platinum-containing regimen or recurrence of disease within 180 days of previous platinum treatment
* Have measurable disease based on modified RECIST 1.1. For the purposes of this study measurable disease is defined at least one "target lesion" that can be accurately measured in at least one dimension (longest dimension to be recorded). Each target lesion must be > 20 mm when measured by conventional techniques, including palpation, plain x-ray, computed tomography (CT), and magnetic resonance imaging (MRI), or > 10 mm when measured by spiral CT. The target lesion must be distinct from other tumor areas selected for pre-treatment biopsies. Pre-treatment imaging must be performed within 4 weeks of starting therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of >= 12 weeks
* Body weight > 30 kg. Note: if subject's weight falls below 30 kg during study but the patient is otherwise eligible to continue investigational therapy the dose of durvalumab will be modified to be weight-based (20 mg/kg for the 1500 mg dose; modification is not required for 1120 mg dose)
* Hemoglobin >= 9.0 g/dL
* Absolute neutrophil count (ANC) > 1500/mm^3
* Platelet count >= 100 x 10^9/L (> 75,000/mm^3)
* Serum bilirubin =< 1.5 x upper limit of normal (ULN)

  * This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase [SGPT]) =< 2.5 x ULN unless liver metastases are present, in which case it must be =< 5 x ULN
* Measured creatinine clearance (CL) > 40 mL/min or calculated creatinine CL > 40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance
* Evidence of post-menopausal status or negative serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy)
  * Women >= 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy)
* Patients must have no currently available standard of care treatment options

Exclusion Criteria:

* Participation in another clinical study with an investigational product (IP) during the last 28 days
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) =< 28 days prior to the first dose of study drug. If sufficient wash-out time has not occurred due to the schedule or pharmacokinetic (PK) properties of an agent, a longer wash-out period will be required, as agreed by AstraZeneca, Aravive, and the investigator
* Any unresolved toxicity National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade >= 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

  * Patients with grade >= 2 neuropathy will be evaluated on a case-by-case basis after consultation with the primary investigator
  * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the study physician
* Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment
* Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable
* History of allogenic organ transplantation
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia;
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement;
  * Any chronic skin condition that does not require systemic therapy;
  * Patients without active disease in the last 5 years may be included but only after consultation with the primary investigator;
  * Patients with celiac disease controlled by diet alone
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring Adverse Events (AEs) or compromise the ability of the patient to give written informed consent
* Any medical, social, or psychological condition that would interfere with evaluation of study treatment or interpretation of patient safety or study results
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis [TB] testing in line with local practice), hepatitis B (known positive hepatitis B virus [HBV] surface antigen [HBsAg] result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA)
* History of another primary malignancy except for the following histories:

  * Malignancy treated with curative intent and with no known active disease >= 5 years before the first dose of IP and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* History of leptomeningeal carcinomatosis
* Brain metastases or spinal cord compression. Patients with suspected brain metastases at screening should have a magnetic resonance imaging (MRI) (preferred) or computed tomography (CT), each preferably with intravenous (IV) contrast of the brain prior to study entry
* Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) >= 470 ms
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or AVB-S6-500. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection);
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent;
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 90 days after the last dose of IP
* Female patients who are pregnant or breastfeeding or of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab + AVB-S6-500 combination therapy
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients
* Unresolved partial or complete small or large bowel obstruction
* Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir A Jazaeri, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruitment was from December 2019 until November 2022 and all recruitments were done in a medical clinic setting.
Groups:
- Phase 1: Durvalumab 1500 mg IV every 4 weeks + AVB-S6-500 10 mg/kg IV every 2 weeks
- Phase 2A: Monotherapy with AVB-S6-500 IV 10 mg/kg every 2 weeks for 6 weeks then combination of Durvalumab 1500 mg IV every 4 weeks + AVB-S6-500 10 mg/kg IV every 2 weeks
- Phase 2D: Monotherapy with Durvalumab 1500 mg IV every 4 weeks for 6 weeks then combination of Durvalumab 1500 mg IV every 4 weeks + AVB-S6-500 10 mg/kg IV every 2 weeks
Period: Overall Study
Arm/Group | Phase 1 | Phase 2A | Phase 2D
Started | 11 | 0 | 0
Completed | 10 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated early due to sponsor closing the study. The study never progressed passed phase 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 | Phase 2A | Phase 2D | Total
Number analyzed (Participants) | 11 | 0 | 0 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  | 0
  Between 18 and 65 years | 10 |  |  | 10
  >=65 years | 1 |  |  | 1
Age, Continuous [Mean (Full Range); unit: years] | 56.9 [45 to 73] |  |  | 56.9 [45 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 |  |  | 11
  Male | 0 |  |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 |  |  | 2
  Not Hispanic or Latino | 9 |  |  | 9
  Unknown or Not Reported | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0
  Asian | 1 |  |  | 1
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 0 |  |  | 0
  White | 8 |  |  | 8
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 2 |  |  | 2
Region of Enrollment [Number; unit: participants]
  United States | 11 |  |  | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Time Frame: 35 months
Population: Treatment never progressed passed phase 1.
Measure: Number; unit: participants
Arm/Group | Phase 1 | Phase 2A | Phase 2D
Number analyzed (Participants) | 11 | 0 | 0
participants
  Grade 1 AEs | 11 |  |
  Grade 2 AEs | 9 |  |
  Grade 3 AEs | 3 |  |
  Grade 2 SAEs | 2 |  |
  Grade 3 SAEs | 1 |  |

2. Secondary Outcome: To Estimate Objective Response Rate to Combination AVB-S6-500 and Durvalumab Therapy
Time Frame: 35 months
Population: Treatment never progressed passed phase 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 | Phase 2A | Phase 2D
Number analyzed (Participants) | 11 | 0 | 0
Participants | 11 |  |

3. Secondary Outcome: To Estimate the Median Immune-related Progression Free Survival (irPFS) as Well as Overall Survival OS by RECIST 1.1 After Treatment With Combination Durvalumab and AVB-S6-500
Time Frame: 35 months
Population: Treatment never progressed passed phase 1.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1 | Phase 2A | Phase 2D
Number analyzed (Participants) | 11 | 0 | 0
Months
  PFS | 1.81 [1.71 to 2.40] |  |
  OS | 4.53 [2.10 to 24.74] |  |

4. Secondary Outcome: To Investigate Molecular and Immunological Changes Associated With the Combination of AVBS6-500 and Durvalumab.
Description: Serum fractions will be isolated from blood samples collected in EDTA-free tubes and will be used to measure GAS6 suppression, which will be analyzed by Altasciences.
Time Frame: 35 months
Population: Treatment never progressed passed phase 1.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Phase 1 | Phase 2A | Phase 2D
Number analyzed (Participants) | 11 | 0 | 0
ng/mL | 30.5 [5.6 to 45.1] |  |

ADVERSE EVENTS:
Time Frame: 35 months
Description: NCI CTCAE version 4.03
Arm/Group | Phase 1 | Phase 2A | Phase 2D
All-Cause Mortality (participants affected / at risk) | 1/11 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 3/11 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 11/11 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 (N=11) | Phase 2A (N=0) | Phase 2D (N=0)
Infusion related reaction (General disorders) | 2 (3) | 0 | 0
Lung Infection (Infections and infestations) | 1 (1) | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 (N=11) | Phase 2A (N=0) | Phase 2D (N=0)
Anemia (Blood and lymphatic system disorders) | 2 (5) | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 (1) | NA | NA
Alkaline phosphatase increased (Investigations) | 1 (1) | NA | NA
Anorexia (Metabolism and nutrition disorders) | 2 (2) | NA | NA
Aspartate aminotransferase increased (Investigations) | 3 (3) | NA | NA
Bloating (Gastrointestinal disorders) | 1 (1) | NA | NA
Constipation (Gastrointestinal disorders) | 4 (5) | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | NA
Creatinine increased (Investigations) | 3 (3) | NA | NA
Diarrhea (Gastrointestinal disorders) | 1 (1) | NA | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | NA | NA
Fatigue (General disorders) | 3 (4) | NA | NA
Headache (Nervous system disorders) | 1 (1) | NA | NA
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | NA | NA
Hyperparathyroidism (Endocrine disorders) | 1 (1) | NA | NA
Hypertension (Vascular disorders) | 1 (1) | NA | NA
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | NA | NA
Hyponatremia (Metabolism and nutrition disorders) | 3 (4) | NA | NA
Infusion related reaction (General disorders) | 1 (1) | NA | NA
Investigations - Other, TSH decreased (Investigations) | 1 (1) | NA | NA
Investigations - Other, GGT increased (Investigations) | 1 (1) | NA | NA
Lipase increased (Investigations) | 1 (1) | NA | NA
Lung infection (Infections and infestations) | 1 (1) | NA | NA
Lymphocyte count decreased (Investigations) | 1 (1) | NA | NA
Nausea (Gastrointestinal disorders) | 5 (6) | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | NA | NA
Serum amylase increased (Investigations) | 2 (3) | NA | NA
Tremor (Nervous system disorders) | 1 (1) | NA | NA
Vomiting (Gastrointestinal disorders) | 3 (5) | NA | NA
White blood cell decreased (Investigations) | 1 (1) | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT04019288/Prot_SAP_001.pdf
  • Informed Consent Form (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT04019288/ICF_000.pdf